CLINICAL TRIAL: NCT04545866
Title: Randomized Controlled Trial of Budesonide + Surfactant Versus Surfactant Alone in Extremely Preterm Infants ("The Budesonide in Babies (BiB) Trial")
Brief Title: The Budesonide in Babies (BiB) Trial
Acronym: BiB
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NICHD-NRN-0064; UG1HD034216 (NIH); UG1HD027904 (NIH); UG1HD021364 (NIH); UG1HD027853 (NIH); UG1HD040689 (NIH); UG1HD040492 (NIH); UG1HD027851 (NIH); UG1HD087229 (NIH); UG1HD053109 (NIH); UG1HD068278 (NIH); UG1HD068244 (NIH); UG1HD068263 (NIH); UG1HD027880 (NIH); UG1HD053089 (NIH); UG1HD087226 (NIH); UG1HD112079 (NIH); UG1HD112097 (NIH); UG1HD112100 (NIH); 3U24HD095254-07 (NIH)
Record Dates: First submitted 2020-09-04; First posted 2020-09-11 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Bronchopulmonary Dysplasia (BPD); Respiratory Distress Syndrome; Prematurity; Extreme; Neonatal
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Respiratory Distress Syndrome; Premature Birth | interventions — Budesonide; Surface-Active Agents; poractant alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigator, primary providers, primary data collectors, and participants will be masked to randomization arm assignment. Only research pharmacists and a designated respiratory therapist (or other qualified person) will be unmasked at the enrolling sites. The designated respiratory therapist (or other qualified person) must be unmasked to allow drug mixing at bedside for expeditious study drug administration; however, this person will not be the primary medical provider nor the primary data collector for that infant, and will not be otherwise involved in the research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- budesonide with surfactant (Experimental): Infants randomized to the intervention arm receive a dose of surfactant (poractant alfa; Curosurf) mixed with budesonide (Pulmicort nebulizing suspension) within 50 hours of birth and administered via endotracheal tube.
  Interventions: Drug: budesonide (Pulmicort nebulizing suspension).
- surfactant alone (Active Comparator): Infants randomized to the active control arm receive a dose of surfactant (poractant alfa; Curosurf).
  Interventions: Drug: surfactant (poractant alfa;Curosurf)

INTERVENTIONS:
Drug: budesonide (Pulmicort nebulizing suspension). — The first dose of budesonide is 0.25 mg/kg in a volume of 1 ml/kg, for a total volume of 2.5 ml/kg of Curosurf + 1 ml/kg of budesonide. If the infant is to receive a second dose of study drug within 50 hours of birth, the dosage of Curosurf is 1.25 ml/kg for the second dose and 1 ml/kg of budesonide.
  Other Names: Pulmicort nebulizing suspension.
  Arms: budesonide with surfactant
Drug: surfactant (poractant alfa;Curosurf) — The first dose of surfactant (poractant alfa; Curosurf) is 2.5 ml/kg. If the infant is to receive a second dose of study drug within 50 hours of birth, the dosage of Curosurf is 1.25 ml/kg for the second dose.
  Other Names: poractant alfa;Curosurf
  Arms: surfactant alone

SUMMARY:
This is a Phase 3, randomized, masked, active-controlled, multicenter trial designed to determine whether early intratracheal administration of a combination of budesonide with surfactant, as compared to surfactant alone, will reduce the incidence of physiologic bronchopulmonary dysplasia (BPD) or death by 36 weeks' post-menstrual age in extremely preterm infants.

DETAILED DESCRIPTION:
From a study of 9575 extremely preterm (22-28 weeks gestational age and 401-1500g birth weight) infants born between 2003 and 2007 and enrolled in the Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Neonatal Research Network (NRN), it is anticipated that 93% of extremely preterm infants will develop respiratory distress syndrome, 68% will develop bronchopulmonary dysplasia (BPD), 16% will develop severe intraventricular hemorrhage, and 36% will develop late-onset sepsis (PMID: 20732945). Furthermore, in 2014 20% of the infants enrolled in the NRN Generic Database (GDB) died (8% by less than 12 hours, 12% between 12 hours and 120 days, and 1% after 120 days) and 47% of infants who survived to 36 weeks' post-menstrual age (PMA) developed physiologic BPD (NRN GDB data). BPD is therefore one of the most common morbidities in extremely preterm infants. Death is a competing outcome for BPD, as infants who die before ascertainment of BPD at 36 weeks' PMA cannot be diagnosed with BPD even though they may have been at the highest risk. As children get older, BPD has been shown to be associated with worse cognitive outcomes in school age and with abnormal pulmonary function in adolescence and adulthood (PMID: 14595077; 15499947; 2247118).

Recent randomized trials have indicated a lower incidence of BPD/death with the use of a combination of budesonide with surfactant (budesonide + surfactant) compared to surfactant alone when administered soon after birth. Therefore, after obtaining informed consent and confirming eligibility for the trial, infants are randomized in a 1:1 allocation ratio to either the budesonide + surfactant arm or the surfactant alone arm within 48 hours of birth.

ELIGIBILITY:
Inclusion Criteria:

* Liveborn infants 22 0/7 - 28 6/7 weeks gestation or 401 - 1000 grams (inclusive) birth weight
* Clinical decision to give surfactant
* Less than or equal to 48 hours postnatal age

Exclusion Criteria:

* Terminal illness (heart rate < 100 beats per minute, unresponsiveness to resuscitation) or unlikely to survive as judged by the clinician
* Decision to redirect or limit support
* Use of surfactant before enrollment (first dose of surfactant must be study drug)
* Infant received systemic steroids prior to enrollment
* Use of indomethacin, either received by the mother within 24 hours prior to delivery,received by the infant prior to enrollment, or intent to administer to the infant for IVH prophylaxis or PDA management from enrollment up to 7 days of final dose of study drug
* Serious chromosomal abnormalities or major malformations
* Known congenital infections including, but not limited to, confirmed sepsis, congenital CMV, etc.
* Infants with a permanent neuromuscular condition that affects respiration
* Enrollment in a conflicting clinical trial

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 642 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2026-12-17 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Namasivayam Ambalavanan, MD, Principal Investigator — University of Alabama at Birmingham
Locations (19):
- United States (19):
  - University of Alabama, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Sharp Mary Birch Hospital for Women & Newborns, San Diego, California
  - Emory University, Atlanta, Georgia
  - Northwestern Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Mississippi Medical Center - Children's of Mississippi, Jackson, Mississippi
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Brown University - Women and Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
NIH has had a long-standing policy to share and make available to the public the results and accomplishments of the activities that it funds. The NRN plans to share de-identified data after final publication in an NIH supported data repository such as the NICHD Data and Specimen Hub (https://dash.nichd.nih.gov).

REFERENCES:
- [Derived] Ambalavanan N, Carlo WA, Nowak KJ, Wiener LE, Cosby SS, Bhatt AJ, Watterberg KL, Poindexter BB, Keszler M, D'Angio CT, Brion LP, Narendran V, Rau CA, Cotten CM, Laughon MM, Das A, Rysavy MA, Hibbs AM, Fuller J, Puopolo KM, Katheria A, Patel RM, Bermick JR, Laptook AR, Prelipcean I, Wyckoff MH, Moore R, Merhar SL, Ohls RK, Yoder BA, Perez M, Ghavam S, Meyer LR, Chock VY, DeMauro SB, Jackson WM, Handa D, Walsh MC; National Institute of Child Health and Human Development Neonatal Research Network. Early Intratracheal Budesonide to Reduce Bronchopulmonary Dysplasia in Extremely Preterm Infants: The Budesonide in Babies (BiB) Randomized Clinical Trial. JAMA. 2025 Oct 28;334(16):1452-1462. doi: 10.1001/jama.2025.16450. PMID 41026481

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One infant was randomized and treated in error after the parent/guardian declined consent. The infant was withdrawn from the trial upon discovery of the protocol violation. At the parent's request, the infant's data have been fully redacted. No data are available for reporting or analysis (including treatment allocation), and this participant is excluded from the intention to treat (ITT) population.
Groups:
- Budesonide + Surfactant: Budesonide (Pulmicort nebulizing suspension) 1 ml/kg + Surfactant (poractant alfa; Curosurf) 2.5 ml/kg
- Surfactant Alone: Surfactant (poractant alfa; Curosurf) 2.5 ml/kg
Period: Overall Study
Arm/Group | Budesonide + Surfactant | Surfactant Alone
Started | 323 | 318
Completed (Completed Study) | 321 | 318
Not Completed | 2 | 0
Not completed — Withdrawal by Parent(s)/Legal Guardian(s) | 1 | 0
Not completed — Withdrawal by Physician | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- BUDE: Budesonide (Pulmicort nebulizing suspension) 1 ml/kg + Surfactant (poractant alfa; Curosurf) 2.5 ml/kg
- SURF: Surfactant (poractant alfa; Curosurf) 2.5 ml/kg
- Total: Total of all reporting groups
Arm/Group | BUDE | SURF | Total
Number analyzed (Participants) | 323 | 318 | 641
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 25.8 (1.9) | 25.9 (2) | 25.9 (1.9)
Age, Customized [Count of Participants; unit: Participants]
  Greater Than or Equal to 26 0/7 weeks | 185 | 188 | 373
  Less Than 26 0/7 weeks | 138 | 130 | 268
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 163 | 156 | 319
  Male | 158 | 162 | 320
  Missing | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African America | 101 | 122 | 223
  Other | 21 | 17 | 38
  Unknown or Not Reported | 18 | 11 | 29
  White | 183 | 168 | 351
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 50 | 54 | 104
  Not Hispanic or Latino | 254 | 254 | 508
  Unknown or Not Reported | 19 | 10 | 29

OUTCOME MEASURES:

1. Primary Outcome: Physiologic BPD or Death by 36 Weeks PMA
Description: A composite outcome for infants who were diagnosed with physiologic BPD or died by 36 weeks PMA. Physiologic BPD is determined using existing NRN GDB criteria at 36 weeks' PMA. Infants alive an in hospital are classified based on respiratory status at 36 week's PMA or by a room air weaning challenge performed between 36 and 37 weeks' PMA. Infants who are transferred or discharged before 36 weeks are classified based on the support they are receiving at that time. Infants who died before 36 weeks' PMA are not assessed for BPD. Deaths include all-cause deaths between randomization and 36 weeks' PMA.
Time Frame: Randomization to 36 weeks PMA
Population: An intent-to-treat (ITT) analysis which included all infants participants who were randomized and who provided outcome data.
Measure: Count of Participants; unit: Participants
Arm/Group | BUDE | SURF
Number analyzed (Participants) | 323 | 318
Participants
  No | 101 | 102
  Unknown | 2 | 0
  Yes | 220 | 216

2. Secondary Outcome: Death by 36 Weeks PMA
Description: Died (all-cause) after randomization and by 36 weeks PMA
Time Frame: Randomization to 36 weeks PMA
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BUDE | SURF
Number analyzed (Participants) | 323 | 318
Participants
  No | 272 | 276
  Unknown | 2 | 0
  Yes | 49 | 42

3. Secondary Outcome: Physiologic BPD
Description: Diagnosed with physiologic BPD at 36 weeks PMA. Physiologic BPD is determined using existing NRN GDB criteria at 36 weeks' PMA. Infants alive an in hospital are classified based on respiratory status at 36 week's PMA or by a room air weaning challenge performed between 36 and 37 weeks' PMA. Infants who are transferred or discharged before 36 weeks are classified based on the support they are receiving at that time. Infants who died before 36 weeks' PMA are not assessed for BPD.
Time Frame: At 36 weeks PMA
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BUDE | SURF
Number analyzed (Participants) | 323 | 318
Participants
  No | 101 | 102
  Unknown | 51 | 42
  Yes | 171 | 174

4. Secondary Outcome: Grade of BPD Severity
Description: BPD Severity Grade at 36 weeks PMA according to the Jensen et al. (2019; PMID: 30995069) definition, also known as pragmatic BPD. Infants are assess based on the mode of support at 36 weeks' postmenstrual age regardless of prior duration or current level of oxygen therapy.
Time Frame: At 36 weeks PMA
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BUDE | SURF
Number analyzed (Participants) | 323 | 318
Participants
  Grade 0 (No BPD) | 70 | 66
  Grade 1 (Mild BPD) | 72 | 78
  Grade 2 (Moderate BPD) | 99 | 100
  Grade 3 (Severe BPD) | 28 | 26
  Unknown | 54 | 48

5. Secondary Outcome: Severe BPD
Description: Diagnosed with Severe (Grade 3) BPD at 36 weeks PMA according to the Jensen et al. (2019; PMID: 30995069) definition. This outcome is a dichotomy of the pragmatic BPD severity grades (Grade 3 vs. Grade 2, 1, or 0).
Time Frame: At 36 weeks PMA
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BUDE | SURF
Number analyzed (Participants) | 323 | 318
Participants
  No | 241 | 244
  Unknown | 54 | 48
  Yes | 28 | 26

6. Secondary Outcome: Use of Additional Postnatal Steroids
Description: Use of any postnatal steroids for treatment of evolving chronic lung disease (separate from study drug) between 7 days after the final dose of study drug and 36 weeks PMA.
  Note: Infants were permitted up to two doses of study drug within 50 hours postnatal age, so this outcome spans 7-10 days postnatal age through 36 weeks postmenstrual age.
Time Frame: 7 days post last dose of study drug through 36 weeks PMA
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BUDE | SURF
Number analyzed (Participants) | 323 | 318
Participants
  No | 216 | 202
  Unknown | 5 | 7
  Yes | 102 | 109

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from treatment through 7 days (168 hours) post-treatment, or treatment through 30 days (720 hours) post-treatment for SIP and PVL. All-cause mortality was monitored from randomization through 36 weeks PMA.
Description: AE onset was monitored from treatment initiation through 7 days after the last dose of study drug (30 days for SIP and PVL). This window includes up to 10 days postnatal age (or 33 days PNA for SIP/PVL). AEs were not monitored for infants who did not initiate treatment.
  All-cause mortality was monitored from randomization through 36 weeks PMA or prior study status (discharge, transfer).
  Note: Treatment group is reported as randomized. Published analyses may use treatment as received.
Arm/Group | BUDE | SURF
All-Cause Mortality (participants affected / at risk) | 49/323 | 42/318
Serious Adverse Events (participants affected / at risk) | 63/323 | 55/318
Other Adverse Events (participants affected / at risk) | 232/323 | 187/318
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BUDE (N=323) | SURF (N=318)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest neonatal (Cardiac disorders) | 0 (0) | 1 (1)
Newborn persistent pulmonary hypertension (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Pulmonary hypoplasia (Congenital, familial and genetic disorders) | 1 (1) | 2 (2)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 14 (14) | 6 (6)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Necrotising colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neonatal intestinal perforation (Gastrointestinal disorders) | 0 (0) | 4 (4)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 6 (6) | 2 (2)
Sepsis neonatal (Infections and infestations) | 2 (2) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (8) | 3 (3)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 15 (15) | 17 (17)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Intraventricular haemorrhage neonatal (Nervous system disorders) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Neonatal pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Pulmonary air leakage (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 8 (8)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary hypertensive crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 13 (14) | 7 (7)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BUDE (N=323) | SURF (N=318)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Newborn persistent pulmonary hypertension (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Necrotising colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Necrotising enterocolitis neonatal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 6 (6) | 5 (5)
Sepsis neonatal (Infections and infestations) | 5 (5) | 3 (3)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperammonaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 208 (263) | 154 (191)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 20 (20) | 17 (17)
Intraventricular haemorrhage neonatal (Nervous system disorders) | 3 (3) | 1 (1)
Periventricular leukomalacia (Nervous system disorders) | 5 (5) | 2 (2)
Device occlusion (Product Issues) | 1 (1) | 3 (3)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Pulmonary air leakage (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Pulmonary haemorrhage neonatal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary interstitial emphysema syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Hypertension (Vascular disorders) | 28 (31) | 20 (22)
Hypotension (Vascular disorders) | 42 (45) | 53 (57)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-09-08): https://cdn.clinicaltrials.gov/large-docs/66/NCT04545866/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-10): https://cdn.clinicaltrials.gov/large-docs/66/NCT04545866/SAP_001.pdf